CLINICAL TRIAL: NCT07139691
Title: Efficacy of TAP Block in Postoperative Pain Management for Elective Hysterectomy: a Randomized Controlled Clinical Trial
Brief Title: TAP Block With Lidocaine and Ropivacaine 0.2% (0.4 ml/kg/Side) for Pain and Opioid Reduction After Hysterectomy
Acronym: TAP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Matild Keresztes (Other)
Responsible Party: Sponsor-Investigator, Matild Keresztes, Doctor, Tîrgu Mureș Emergency Clinical County Hospital, Romania
Organization: Tîrgu Mureș Emergency Clinical County Hospital, Romania (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 651/12.01.2024
Record Dates: First submitted 2025-07-29; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Postoperative Pain Following Hysterectomy
Keywords: Transversus Abdominis Plane Block; Postoperative Pain Management; Hysterectomy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: TAP Block with Lidocaine and Ropivacaine (Experimental): Participants in this arm will receive a pre-incisional Transversus Abdominis Plane (TAP) block performed under ultrasound guidance. The block will be administered bilaterally using a mixture of lidocaine and ropivacaine 0.2% with a calculated dose of 0.4 ml/kg per side, in addition to standard analgesia.
  Interventions: Procedure: Pre-incisional Transversus Abdominis Plane (TAP) block performed under ultrasound guidance. The block will be administered bilaterally using a mixture of lidocaine and ropivacaine 0.2%
- Arm 2: Standard Analgesia (Control) (Active Comparator): Participants in this arm will receive standard analgesia for postoperative pain management following elective hysterectomy. This regimen typically includes systemic analgesics (e.g., intravenous or oral non-opioid analgesics and opioids as needed) but does not include a Transversus Abdominis Plane (TAP) block.
  Interventions: Drug: Participants in this arm will receive standard analgesia for postoperative pain management following elective hysterectomy

INTERVENTIONS:
Procedure: Pre-incisional Transversus Abdominis Plane (TAP) block performed under ultrasound guidance. The block will be administered bilaterally using a mixture of lidocaine and ropivacaine 0.2% — After the induction of general anesthesia, bilateral TAP block will be performed in patients from Group 1. The administered dose will include 0.2% lidocaine combined with 0.2% ropivacaine, at a dose of 0.4 ml/kg per side, without exceeding toxic dose limits per kg.
  Arms: Arm 1: TAP Block with Lidocaine and Ropivacaine
Drug: Participants in this arm will receive standard analgesia for postoperative pain management following elective hysterectomy — Participants in this arm will receive standard multimodal systemic analgesia for postoperative pain management following elective hysterectomy. The regimen includes Paracetamol (oral or intravenous) 1g/24 hour, Ibuprofen IV 1200 mg/24 hour, or Parecoxib 80 mg/24 hour IV, and Tramadol 100 mg IV. Additional rescue doses of Tramadol (50-100 mg IV every 4-6 hours) may be administered based on pain intensity, with a maximum of 400 mg/24 hours (or 300 mg/24 hours for patients aged ≥75 years). No Transversus Abdominis Plane (TAP) block will be performed in this group. Pain intensity, opioid use, and postoperative recovery scores will be evaluated and compared with the TAP block intervention group.
  Arms: Arm 2: Standard Analgesia (Control)

SUMMARY:
The goal of this study is to evaluate whether the Transversus Abdominis Plane (TAP) block can effectively reduce postoperative pain and opioid consumption in patients undergoing elective hysterectomy.

The main questions it aims to answer are:

Primary outcome: Does performing a pre-incisional TAP block reduce postoperative pain scores and opioid consumption compared to standard analgesic management?

Secondary outcomes:

Does TAP block reduce intraoperative opioid requirements during hysterectomy? Does TAP block enhance postoperative recovery and facilitate early mobilization? Does TAP block reduce the length of hospital stay? Does TAP block improve overall patient satisfaction following hysterectomy? If there is a comparison group: Researchers will compare patients receiving TAP block with lidocaine and ropivacaine (0.2%, 0.4 ml/kg per side) to patients receiving standard analgesia without TAP block to see if the TAP block provides superior pain relief, lowers opioid needs, and improves recovery outcomes.

Participants will:

Undergo elective total or subtotal hysterectomy. Receive either a TAP block (intervention group) or standard analgesic management (control group).

Have their intraoperative and postoperative opioid consumption, pain scores, recovery parameters, and satisfaction assessed.

DETAILED DESCRIPTION:
Hysterectomy is a common gynecological surgical procedure involving the removal of the uterus. The procedure may be total or subtotal, and is frequently associated with moderate to severe postoperative pain. Effective management of this pain is crucial and is typically achieved through multimodal analgesia. This approach includes regional nerve blocks, systemic analgesics (oral and intravenous), and adjunctive therapies (physical or psychological), resulting in reduced opioid requirements, minimized side effects, and shorter hospital stays.

The transversus abdominis plane (TAP) block is a regional anesthesia technique involving the injection of a local anesthetic between the transversus abdominis and internal oblique muscles. This targets the thoracolumbar nerves (T6-L1) and provides effective analgesia for the anterior abdominal wall. When performed under ultrasound guidance following abdominal surgery, the TAP block has demonstrated benefits including decreased incisional pain, reduced opioid consumption, and improved postoperative mobilization.

This is a prospective, randomized, comparative clinical trial conducted within the Department of Obstetrics and Gynecology at Mureș County Emergency Clinical Hospital. The study period extends from January 2024 to December 2025 or until the target sample size is reached. All anesthetic and surgical interventions utilized are within standard clinical practice; no experimental drugs or procedures are employed.

The study compares two multimodal analgesia protocols to identify the most effective and satisfactory method of postoperative pain management. All participants will provide written informed consent prior to enrollment.

Participants will be randomly allocated into two groups using a computer-generated randomization application on the day of surgery. The anesthesiologist performing the TAP block will be the only staff member aware of group allocation.

To maintain blinding, all participants will leave the operating room with bilateral lateral abdominal dressings, regardless of group assignment. Postoperative evaluators will be blinded to group allocation.

The transversus abdominis plane (TAP) block will be performed under ultrasound guidance using a Sonosite ultrasound system equipped with a linear probe (6-15 MHz). The block will be executed after induction of general anesthesia, utilizing the lateral approach.

The procedure begins by positioning the ultrasound probe at the level of the umbilicus, oriented transversely to identify the rectus abdominis muscle. The probe is then moved laterally and slightly posteriorly to visualize the three muscle layers of the lateral abdominal wall in cross-section: External oblique, Internal oblique, Transversus abdominis.

The final probe position will be between the iliac crest and the costal margin, where the muscle layers are clearly visualized. Under direct ultrasound visualization, the needle (Stimuplex Ultra 360, 20G × 6, 30° bevel, 100-150 mm) is inserted in-plane, from medial to lateral, puncturing the skin above the probe and advancing through the tissue under the ultrasound beam.

The needle is advanced until it reaches the fascial plane between the internal oblique and transversus abdominis muscles. Correct placement is confirmed by the appearance of the "unzipping" or hydro-dissection effect upon injection of a small volume of local anesthetic, indicating separation of the fascial layers.

The local anesthetic solution is then injected in increments of 5 ml per side, with aspiration performed after each increment to exclude intravascular needle placement.

The entire TAP block procedure is conducted under strict aseptic conditions, including:

* Skin disinfection with Braunol iodine solution
* Use of sterile gloves
* Use of a sterile ultrasound probe cover
* Sterile handling of all equipment and medications Preoperative data collected will include age, weight, height, body mass index (BMI), ASA score, comorbidities, gynecologic diagnosis, and baseline Quality of Recovery score (QoR-15).

Intraoperative data will include: time of anesthesia induction, time of TAP block (if applicable), time of surgical incision, total surgery duration, opioid consumption, heart rate and blood pressure.

Intraoperative pain will be defined as a ≥20% increase in heart rate and/or blood pressure compared to baseline values recorded one day prior to surgery.

Postoperative assessments will include:

* Pain intensity at 0, 1, 4, 6, and 24 hours (at rest and during movement)
* Numeric Rating Scale (0-10)
* Patient satisfaction score at 24 hours
* QoR-15 score at 48 hours Data will be recorded using standardized intraoperative and postoperative forms. The intraoperative form will be completed by the anesthesiologist performing the surgery. The postoperative form will be completed by a blinded evaluator (resident or specialist from another unit). All data will be entered into Microsoft Excel and analyzed using GraphPad Prism.

Results will be statistically analyzed and interpreted to identify differences in pain control, opioid consumption, recovery, and patient satisfaction between the two groups. Conclusions will guide the development of updated institutional pain management protocols for hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery
* Subumbilical incision (median, Phannenstil)
* Total or subtotal hysterectomy
* Age over 18 years

Exclusion Criteria:

* Patient refusal
* Infection at the puncture site
* Chronic pain
* Chronic use of analgesics
* Contraindications to NSAIDs, local anesthetics, or opioids (e.g., tramadol: antidepressants, epileptic disorders)
* Severe hepatic disease
* Renal insufficiency (Creatinine Clearance ≤ 30 ml/min)
* Coagulopathy (Platelet count ≤ 75,000, INR ≥ 1.4)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only biologically female patients are eligible to participate, as hysterectomy is a surgical procedure performed exclusively on individuals with a uterus.
Enrollment: 82 (Estimated)
Dates: Start 2024-01-12 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative Opioid Consumption (Tramadol) | From end of surgery (arrival in recovery room) to 24 hours postoperatively
  Total intravenous Tramadol administered for postoperative pain management will be recorded during the first 24 hours following elective hysterectomy. Unit of Measure: Milligrams (mg) of IV Tramadol
Postoperative Pain Intensity | From end of surgery to 24 hours postoperatively
  Pain intensity will be assessed using the Numeric Rating Scale (NRS), ranging from 0 (no pain) to 10 (worst imaginable pain). Scores will be recorded at 0, 1, 4, 6, and 24 hours postoperatively, both at rest and during movement.

SECONDARY OUTCOMES:
Intraoperative Opioid Consumption During Hysterectomy | From induction of anesthesia until completion of surgery
  Total amount of opioids administered intraoperatively will be recorded. The outcome will assess whether performing a pre-incisional bilateral TAP block reduces opioid requirements during the surgical procedure compared to standard multimodal analgesia alone.
Postoperative Quality of Recovery Assessed by QoR-15 | At 48 hours after completion of surgery
  The Quality of Recovery-15 (QoR-15) questionnaire will be used to evaluate postoperative recovery in patients undergoing elective hysterectomy. QoR-15 is a validated tool that assesses multiple domains of recovery including physical comfort, pain, physical independence, psychological support, and emotional state. Scores range from 0 to 150, with higher scores indicating better recovery. The study will assess whether a pre-incisional bilateral TAP block improves QoR-15 scores compared to standard multimodal analgesia.
Length of Hospital Stay | Up to 2 weeks
  The total duration of hospitalization from the end of surgery until patient discharge. This outcome will evaluate whether a pre-incisional bilateral TAP block reduces the length of hospital stay compared to standard multimodal analgesia in patients undergoing elective hysterectomy.
Patient Satisfaction with Postoperative Pain Management | At 24 hours after completion of surgery
  Patient satisfaction with postoperative pain management will be assessed using a 10-item Patient Satisfaction Questionnaire. Each item consists of a statement regarding the participant's experience with pain control, and responses are provided on a 5-point Likert scale:
  1. = Strongly Disagree
  2. = Disagree
  3. = Neutral
  4. = Agree
  5. = Strongly Agree The total score is calculated by summing the responses to all 10 items. The minimum total score is 10, and the maximum total score is 50, with higher scores indicating greater satisfaction. This outcome will evaluate whether the addition of a pre-incisional bilateral TAP block improves patient satisfaction compared to standard multimodal analgesia.

CONTACTS AND LOCATIONS:
Overall Officials: Janos Szederjesi, MD, PhD, Study Chair — Dept. of Anesthesiology & Intensive Care, George Emil Palade Univ. of Medicine & Pharmacy, Târgu Mureș; Matild Keresztes, MD, Principal Investigator — Dept. of Anesthesiology & Intensive Care, George Emil Palade Univ. of Medicine & Pharmacy, Târgu Mureș
Locations (1):
- County Emergency Clinical Hospital of Targu Mureș, Târgu Mureş, Mureș County, Romania

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the results of this study will be made available to other researchers upon reasonable request for secondary analyses, following publication of the primary results. Access will be granted through a secure data-sharing agreement.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 6 months after primary publication and available for 2 years
Access Criteria: Researchers must submit a methodologically sound proposal that is approved by the study's steering committee. Data will be shared via a secure data repository.